CLINICAL TRIAL: NCT03028961
Title: Randomized Clinical Study Comparing the Effectiveness of the Stanford Letter to the Traditional Advance Directive in Bone Marrow Transplant Recipients
Brief Title: Stanford Letter or Traditional Advance Directive in Advance Care Planning in Patients Undergoing Bone Marrow Transplant
Acronym: BMTSLPRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: BMT313
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Advance Directives; Bone Marrow Transplant
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Stanford Letter, interview) (Experimental): Patients listen to a dialogue on the purpose of ACP. Patients receive a paper copy and online web link to the Stanford Letter and complete and return the form by the day of BMT. After completion of the Stanford Letter, patients undergo a semi-structured, research staff-led interview to evaluate personal perceptions of uncertainty with end-of-life decisions, understanding of the ACP form received, and satisfaction with the ACP form.
  Interventions: Other: Stanford Letter; Other: Interview; Other: Questionnaire Administration
- Group II (traditional advance directive, interview) (Active Comparator): Patients listen to a dialogue on the purpose of ACP. Patients receive a paper copy and online web link to the CA Advance Health Care Directive Form and complete and return the form by the day of BMT. After completion of the CA Advance Health Care Directive Form, patients undergo interview as in Group I.
  Interventions: Other: Interview; Other: Questionnaire Administration; Other: CA Advance Health Care Directive Form

INTERVENTIONS:
Other: Stanford Letter — Receive and complete the Stanford Letter
  Other Names: Communication Intervention
  Arms: Group I (Stanford Letter, interview)
Other: Interview — Undergo semi-structured, research staff-led interview
Other: Questionnaire Administration — Ancillary studies
Other: CA Advance Health Care Directive Form — Receive and complete the CA Advance Health Care Directive Form
  Other Names: Communication Intervention
  Arms: Group II (traditional advance directive, interview)

SUMMARY:
The purpose of the proposed research study is to evaluate whether bone marrow transplant patients prefer the Stanford letter advance care planning tool to the standard Advance directive.

Completion of advance care planning prior to BMT is very important, but not often done. The investigators believe that the Stanford Letter will be preferred by patients and will allow them to feel more comfortable and share more of their wishes with family members and the medical team.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. To compare advance care planning (ACP) completion rate amongst bone marrow transplant (BMT) recipients receiving the Stanford Letter versus the traditional advance directive (AD) through a prospective, pilot randomized controlled trial (RCT).

SECONDARY OBJECTIVES:

I. To evaluate differences in patient preference for choice to prolong life following completion of the ACP tool in each group.

II. To assess uncertainty with decision making regarding end of life care following completion of the ACP tool in each group.

III. To explore patient understanding of and satisfaction with the ACP tool in each group.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (INTERVENTION): Patients listen to a dialogue on the purpose of ACP. Patients receive a paper copy and online web link to the Stanford Letter and complete and return the form by the day of BMT. After completion of the Stanford Letter, patients undergo a semi-structured, research staff-led interview to evaluate personal perceptions of uncertainty with end-of-life decisions, understanding of the ACP form received, and satisfaction with the ACP form.

GROUP II (CONTROL): Patients listen to a dialogue on the purpose of ACP. Patients receive a paper copy and online web link to the California (CA) Advance Health Care Directive Form and complete and return the form by the day of BMT. After completion of the CA Advance Health Care Directive Form, patients undergo interview as in Group I.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* All BMT patients at Stanford who are adults and give consent

Exclusion Criteria:

* Less than 18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
ACP completion rate defined as a completed Advance Directive tool (either Stanford Letter or standard CA AD) brought to Stanford University for upload into the medical record | Up to BMT day 0
  The chi-square (X^2) test will be used to determine a significant difference in proportion of ACP tool completion and preferences for choice to prolong life between the two groups.

SECONDARY OUTCOMES:
Patient preferences for life sustaining measures measured via answers to the ACP questions related to use of cardiopulmonary resuscitation and use of mechanical intubation | Up to BMT day 0
  The X^2 test will be used to determine a significant difference in proportion of ACP tool completion and preferences for choice to prolong life between the two groups.
Uncertainty with decision making regarding end of life care measured related to the Decisional Conflict Scale (DCS) results | Up to BMT day 0
  Will be measured using the DCS uncertainty sub-scale (score 0-15; higher score indicates greater uncertainty). Scores from each group will be compared by t-tests.
Understanding of the ACP tool measured using qualitative and quantitative data obtained through the semi-structured interview and DCS | within 28 days of ACP completion
  Will be measured using the DCS effective decision-making sub-scale (score 0-15; higher scores indicate 6 less effective decision-making). Likert scores of understanding of the ACP from each group will be summarized and compared by t-tests.
Satisfaction with the ACP tool measured using qualitative and quantitative data obtained through the semi-structured interview and DCS | within 28 days of ACP completion
  Will be measured using the DCS effective decision-making sub-scale (score 0-15; higher scores indicate 6 less effective decision-making). Scores from each group will be compared by t-tests. Likert scores of satisfaction with the ACP will be summarized and compared by group using t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Muffly, MD, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States